CLINICAL TRIAL: NCT07042867
Title: Prospective Multicenter Cohort Study for the Development and Evaluation of Risk Stratification Tools for Lung Cancers and Their Postoperative Recurrences Using Multimodal Clinical, Radiological, Tissue and Longitudinal Biological Phenotyping Among People at Risk of Lung Cancer
Acronym: LUCA-pi COHORT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2024-A02828-39
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer (Diagnosis)
Keywords: lung cancer, lung nodules, prevention, dignosis, low dose scan, biomarkers
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: patients with a nodule or lung mass identified on CT scan, with no indication of an immedi (Other): patients with a nodule or lung mass identified on CT scan, with no indication of an immediate diagnostic workup
  Interventions: Biological: biobanking; Radiation: low dose scan
- Group B: cohort of patients with a nodule or lung mass identified on CT with an indication for biops (Other): cohort of patients with a nodule or lung mass identified on CT with an indication for biopsy or excision surgery
  Interventions: Biological: biobanking; Radiation: low dose scan
- Group C: Individuals with at least one risk factor for lung cancer and no prior lung imaging, but no (Other): Individuals with at least one risk factor for lung cancer and no prior lung imaging, but not eligible for lung cancer screening according to INCa criteria.
  Interventions: Biological: biobanking; Radiation: low dose scan

INTERVENTIONS:
Biological: biobanking — blood draw at each time point
Radiation: low dose scan — low dose lung scan will be performed at each timepoint

SUMMARY:
Interventional study with minimal risks and constraints, involving annual assessment of the prevalence and incidence of lung cancer using low-dose contrast-free thoracic CT scans, immunological, inflammatory, metabolic, blood nucleic acid and digestive microbiota profiles; systematic proposal of smoking cessation for active smokers, or assistance in maintaining cessation This is a prospective validation study of risk stratification tools still under development.

The results of this study will be used to design medical devices (software integrating risk stratification tools), which will then be evaluated as part of subsequent Clinical Investigations.

ELIGIBILITY:
Inclusion Criteria:

Group A:

CI 1- Age > 18 years AND CI2a- Person eligible for screening with a nodule or lung mass with no indication of reassessment by CT scan before the next round of screening, as recommended by the multidisciplinary consultation meeting OR CI2b- Person not eligible for screening with a nodule or lung mass with an indication for reassessment by CT scan without immediate diagnostic workup (PET scan, biopsy, surgery) as determined by the multidisciplinary consultation meeting.

Group B CI1- Age > 18 years AND CI2- Indication for biopsy or surgical excision for diagnostic and therapeutic purposes proposed in a multidisciplinary consultation meeting.

Group C CI1a- Age 40 - 75 and daily smoking for at least 20 years initiated before age 15 OR CI1b- Age 50 - 75 and passive smoking for at least 20 years in a closed environment (family or workplace) OR CI1c- Age 50 - 75 and smoking 10 cig/d for 30 years or 15 cig/d for 25 years or 20 pack-years with no withdrawal period OR

CI1d- Age 50 - 75 and daily smoking for at least 10 years combined with at least one other lung cancer risk factor from among :

* Self-reported daily passive smoking for > 10 years (smokers at home or in enclosed environments)
* Self-reported exposure to a lung carcinogen: Radon, coal smoke, soot, diesel, nickel, beryllium, arsenic, cadmium, asbestos
* 1st-degree family history of lung cancer
* Personal history of tobacco-related disease, including atheromatous cardiovascular disease, COPD or emphysema, cancer not monitored by chest imaging
* weekly use of cannabis (joints) for 10 years

All Groups:

* Have signed an informed consent form
* Affiliated with or benefiting from a social security scheme
* Male or female

Exclusion Criteria:

Goups A and B Contraindication to lung biopsy or thoracic surgery for diagnostic or therapeutic purposes

Group C Eligible for lung cancer screening according to INCa* criteria

* Previous cancer < 5 years (except carcinoma in situ of the uterine cervix, basal cell carcinoma of the skin, non-invasive urothelial carcinoma treated for curative purposes without CT lung surveillance, prostate cancer with undiagnosable PSA)
* Symptoms of lung cancer (involuntary weight loss > 10% of usual weight in 1 year, hemoptysis)
* Known history of pulmonary nodule requiring specialized follow-up
* History of pulmonary fibrosis or pulmonary hypertension
* Active pulmonary parenchymal infection
* Severe cardiac or respiratory insufficiency (rest dyspnea)
* Performance status (WHO) 2, 3 or 4

All Groups

* patient privé de liberté
* patient sous tutelle ou curatelle
* femmes enceintes ou allaitantes
* patient dans l'incapacité d'effectuer le suivi de 30 mois

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the radiomics algorithm for characterizing benign vs. malignant lung lesions. | 30 months

SECONDARY OUTCOMES:
Sensitivity and specificity of minimal biological panel based on markers of inflammation, immunity, blood metabolism and stool metagenomics for characterization of benign vs. malignant lung lesions. | 30 months
Sensitivity and specificity of new biomarkers including specific antibodies and circulating nucleic acids for characterization of benign vs. malignant lung lesions. | 30 months
Sensitivity and specificity of a patho-radiomic-based algorithm quantifying the risk of recurrence of operated lung cancers. | 30 months
Sensitivity and specificity of minimal and novel biomarker panels for the prediction of postoperative lung cancer recurrence. | 30 months
Description of biomarker panels among people not eligible for lung cancer screening. | 30 months
Change over time in biomarkers overall, then in each of the following subgroups: - people undergoing lung cancer surgery - smoking cessation patients - people with an incident diagnosis of lung cancer | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: David Boulate, Professor of Medicine, Principal Investigator — Assistance Publique Hopitaux De Marseille

IPD SHARING:
Plan to Share IPD: Undecided